CLINICAL TRIAL: NCT01663051
Title: Evaluation of the Zilver® Vena™ Venous Stent
Acronym: VIVO EU
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-018
Record Dates: First submitted 2012-08-06; First posted 2012-08-13 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Iliofemoral Venous Outflow Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Stent: Stent
  Interventions: Device: Zilver Vena Venous Stent

INTERVENTIONS:
Device: Zilver Vena Venous Stent — Stenting iliofemoral venous outflow obstruction

SUMMARY:
This prospective, non-randomized, multi-center study is intended to evaluate the Zilver® Vena™ stent in the treatment of symptomatic iliofemoral venous outflow obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic venous outflow obstruction in up to two iliofemoral venous segments (one in each limb), demonstrated by:
* CEAP 'C' ≥ 3, or
* VCSS pain score ≥ 2

Exclusion Criteria:

* < 18 years of age
* Pregnant or planning to become pregnant in the next 12 months
* Planned surgical or interventional procedures (except thrombolysis and thrombectomy in preparation for the procedure or vena cava filter placement prior to stent implantation in patients at high risk for pulmonary embolism) within 30 days prior to or after the study procedure.
* Lesions with intended treatment lengths extending into the inferior vena cava or below the level of the lesser trochanter
* Previous stenting of the target vessel
* Iliofemoral venous segment unsuitable for treatment with available sizes of study devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic iliofemoral venous outflow obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events | 1 month
Patency | 12 months
  Assessed via ultrasound

CONTACTS AND LOCATIONS:
Locations (5):
- Klinikum Arnsberg GmbH, Arnsberg, Germany
- Galway University Hospitals, Galway, Ireland
- Hospital Madrid Monteprincipe, Madrid, Spain
- Kantonsspital Winterthur, Winterthur, Switzerland
- Guy's and St Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Derived] O'Sullivan GJ, Waldron D, Mannion E, Keane M, Donnellan PP. Thrombolysis and iliofemoral vein stent placement in cancer patients with lower extremity swelling attributed to lymphedema. J Vasc Interv Radiol. 2015 Jan;26(1):39-45. doi: 10.1016/j.jvir.2014.10.010. PMID 25541444
- [Derived] O'Sullivan GJ, Sheehan J, Lohan D, McCann-Brown JA. Iliofemoral venous stenting extending into the femoral region: initial clinical experience with the purpose-designed Zilver Vena stent. J Cardiovasc Surg (Torino). 2013 Apr;54(2):255-61. PMID 23558660